CLINICAL TRIAL: NCT01559558
Title: Changes of Pad Weight Results and Urethral Pressure Profiles After Reduction of Cystocele by Vaginal Gauze Packing
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Principal Investigator, National Taiwan University Hospital, Ho-Hsiung Lin, Professor of Department of Obstetrics & Gynecology, National Taiwan University Hospital
Other Study IDs: 201104016RC
Record Dates: First submitted 2012-03-06; First posted 2012-03-21 (Estimated); Last update posted 2012-03-21 (Estimated); Status verified 2012-03

CONDITIONS: Cystocele
MeSH Terms: conditions — Cystocele

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- cystocele
  Interventions: Procedure: vaginal packing

INTERVENTIONS:
Procedure: vaginal packing — vaginal packing after urodynamic studies, and repeat urethral pressure profile

SUMMARY:
The purpose of this study is to retrospectively review the impact of vaginal packing on the urodynamic studies, especially for urethral pressure profiles.

ELIGIBILITY:
Inclusion Criteria:

* patients with >= stage II cystocele and underwent urodynamic studies

Exclusion Criteria:

* patients less than 20 patients

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with >/= stage II cystocle
Sampling Method: Non-Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2012-03; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Changes of pad weight and values of urethral pressure profiles after vaginal gauze packing. | 1 day
  Changes of pad weight and values of urethral pressure profiles between before and after vaginal gauze packing

SECONDARY OUTCOMES:
The rate of anti-incontinence surgery using the criteria of pad weight > 8 gm after vaginal gauze packing as the indication of concomitant anti-incontinence surgery during cystocele repair | 5 years
  The rate of anti-incontinence surgery in the follow-up period after cystocele repair using the criteria of pad weight > 8 gm after vaginal gauze packing in the initial urodynamic examinations as the indication of concomitant anti-incontinence surgery during cystocele repair.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan, Taiwan